CLINICAL TRIAL: NCT06402331
Title: A Phase 2, Randomized, Open-Label, Multicenter Study to Evaluate the Safety and Efficacy of FPI-2265 (225Ac-PSMA-I&T) in Patients With PSMA-Positive Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: FPI-2265 (225Ac-PSMA-I&T) for Patients With PSMA-Positive Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Acronym: AlphaBreak
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fusion Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FPI-2265-202
Record Dates: First submitted 2024-04-26; First posted 2024-05-07 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: mCRPC; 225Ac-PSMA-I&T; Radioligand therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Part A Arm 1 (Experimental)
  Interventions: Drug: FPI-2265
- Part A Arm 2 (Experimental)
  Interventions: Drug: FPI-2265
- Part A Arm 3 (Experimental)
  Interventions: Drug: FPI-2265
- Part B Arm 4 (Experimental): to be utilized based on analysis of Part A
  Interventions: Drug: FPI-2265
- Part B Arm 5 (Experimental): to be utilized based on analysis of Part A
  Interventions: Drug: FPI-2265
- Part B Arm 6 (Experimental)
  Interventions: Drug: FPI-2265
- Part B Arm 7 (Experimental)
  Interventions: Drug: FPI-2265

INTERVENTIONS:
Drug: FPI-2265 — Investigational treatment FPI2265 is a PSMA ligand radiolabelled with 225Ac.
  Other Names:
  225Ac-PSMA-I&T

SUMMARY:
This is an open-label, randomized, multicenter study of FPI-2265 (225Ac-PSMA-I&T). Patient population is adult participants with PSMA positive mCRPC who have had previous treatment with with 177Lu-PSMA-617 or another 177Lu-PSMA radioconjugate (RC). The purpose of the study is to determine the safety and tolerability, and recommended dose and regiment of FPI-2265.

DETAILED DESCRIPTION:
This is an open-label, randomized, multicenter study of FPI-2265 (225Ac-PSMA-I&T). The purpose of this dose optimization study is to determine the recommended FPI-2265 dose and regimen. Conclusions will be based on safety, tolerability, and anti-tumor activity.

Screening Period: At screening, participants will be assessed for eligibility and undergo a positron emission tomography (PET)/computed tomography (CT) scan to evaluate PSMA positivity. Only participants with PSMA positive cancer and confirmed eligibility criteria will be randomized.

Participants randomized will enter the treatment period and receive investigational doses of FPI2265 according to the dose level and schedule as specified per proposed dose arm.

Part A participants will enroll 1:1:1 at three dose level/schedules, to arms 1, 2 or 3

Part B participants will enroll after completion of part A, in a 1:1 randomization scheme to arms 6 or 7.

Once Part A is fully enrolled and participants have been followed for at least 12 weeks, data from Arm 1 and 2 will be analyzed to assess the feasibility of enrolling participants to arms 4 and 5.

All participants will be monitored and assessed for efficacy response, disease progression and adverse events.

Supportive care will be allowed in all arms at the discretion of the investigator and includes available care for the eligible participant according to best institutional practice for mCRPC treatment, including androgen deprivation therapy (ADT).

Follow-up after end of treatment visit will proceed for 5 years.

5 participants will be enrolled into a dosimetry substudy (open at select sites only). Dosimetry substudy participants will be administered one dose at of FPI2265 and proceed with dosimetric assessments will be taken at a number of timepoints after dose administration.

ELIGIBILITY:
Key Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Diagnosis of adenocarcinoma of prostate proven by histopathology.
* Must have had prior orchiectomy and/or ongoing androgen-deprivation therapy and a castrate level of serum/plasma testosterone
* Progressive mCRPC at time of study entry.
* Must have been previously treated with lutetium-PSMA therapy (lutetium-177 vipivotide tetraxetan or other lutetium-177-PSMA RLT). Treatment must have been completed >6 weeks prior to the first dose of study drug.
* Participants with known BRCA mutations should have received FDA-approved therapies such as PARP inhibitors, per Investigator discretion.
* Positive PSMA PET/CT scan
* Adequate organ function
* For participants who have partners of childbearing potential: Partner and/or participant must not be planning to conceive and must use a method of birth control with adequate barrier protection deemed acceptable by the Principal Investigator during the study treatment and for six months after last study drug administration.

Key Exclusion Criteria:

* Participants who received more than two prior lines of cytotoxic chemotherapy for CRPC.
* Participants who progress prior to administration of the 3rd cycle of prior treatment with 177Lu-PSMA therapy
* All prior treatment-related adverse events must have resolved to Grade ≤1 (CTCAE v5.0). Alopecia and stable persistent Grade 2 peripheral neuropathy may be allowed at the discretion of the Investigator.
* Participants with known, unresolved, urinary tract obstruction are excluded.
* Administration of any systemic cytotoxic or investigational therapy ≤30 days of the first dose of study treatment or five half-lives, whichever is shorter. Completion of large-field external beam radiotherapy ≤four weeks of the first dose of study treatment.
* Participants with a history of central nervous system (CNS) metastases are excluded except those who have received therapy
* Participants with any liver metastases will be excluded
* Participants with skeletal metastases presented as a superscan on a ⁹⁹ᵐTc bone scan.
* Previous or concurrent cancer that is distinct from the cancer under investigation in primary site or histology, except treated cutaneous basal cell carcinoma or squamous cell carcinoma and superficial bladder tumors. Any cancer curatively treated >two years prior to the first dose of treatment is permitted.
* Concurrent serious (as determined by the investigator) medical conditions
* Major surgery ≤30 days prior to the first dose of study treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2026-07-23 (Estimated); Study Completion 2031-01-23 (Estimated)

PRIMARY OUTCOMES:
Frequency, duration, and severity of treatment-emergent adverse events (TEAEs) | From first dose until end of long-term follow-up, 5 years from end of treatment visit.
  Frequencies and percentages of participants with TEAEs will be summarized. Analysis will also be completed regarding duration of TEAEs and their severity.
Frequency and proportion of participants with PSA50 response | From first dose until 12 weeks after the first administered dose of FPI-2265.
  PSA50 response is defined as a decline in PSA levels by at least 50% and is used to evaluate anti-tumor activity.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Barnett, Study Director — Fusion Pharmaceuticals Inc.
Locations (18):
- United States (18):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Hoag Health Center Irvine, Irvine, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - UCSF School of Medicine, San Francisco, California
  - Biogenix Molecular, LLC, Miami, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - United Theranostics, Glen Burnie, Maryland
  - BAMF Health, Grand Rapids, Michigan
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - XCancer, Omaha, Nebraska
  - New Mexico Oncology Hematology Consultants Ltd., Albuquerque, New Mexico
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center - NYC, New York, New York
  - Oregon Health and Science University (OHSU, Knight Cancer Center), Portland, Oregon
  - VA North Texas Health Care System, Nuclear Medicine Service, Dallas, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - U.T. MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No